CLINICAL TRIAL: NCT01203501
Title: In Utero Magnesium Sulfate Exposure: Effects on Extremely-Low-Birth-Weight (ELBW) Infants
Brief Title: In Utero Magnesium Sulfate Exposure: Effects on Extremely-Low-Birth-Weight Infants
Acronym: MgSO4
Status: Completed | Type: Observational
Sponsor: NICHD Neonatal Research Network (Network)
Collaborators: National Center for Research Resources (NCRR) (NIH)
Responsible Party: James A. Lemons, Lead Principal Investigator, Indiana University
Other Study IDs: NICHD-NRN-0016; U10HD034216 (NIH); U10HD027904 (NIH); U10HD021364 (NIH); M01RR000080 (NIH); U10HD027853 (NIH); M01RR008084 (NIH); U10HD027851 (NIH); M01RR000039 (NIH); U10HD034167 (NIH); M01RR001032 (NIH); M01RR002635 (NIH); U10HD027856 (NIH); M01RR000750 (NIH); U10HD021397 (NIH); U10HD027881 (NIH); M01RR000997 (NIH); U10HD027880 (NIH); M01RR000070 (NIH); U10HD021415 (NIH); U10HD021373 (NIH); M01RR000633 (NIH); U10HD021385 (NIH); U10HD027871 (NIH); M01RR006022 (NIH)
Record Dates: First submitted 2010-09-15; First posted 2010-09-16 (Estimated); Last update posted 2017-09-26 (Actual); Status verified 2017-09

CONDITIONS: Infant, Newborn; Infant, Low Birth Weight; Infant, Small for Gestational Age; Infant, Premature; Intracranial Hemorrhages; Leukomalacia, Periventricular; Cerebral Palsy
Keywords: NICHD Neonatal Research Network; Extremely Low Birth Weight (ELBW); Prematurity; Antenatal Magnesium sulfate
MeSH Terms: conditions — Premature Birth; Intracranial Hemorrhages; Leukomalacia, Periventricular; Cerebral Palsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study examined the effect of magnesium sulfate (MgSO4) exposure on adverse outcome in extremely low birth weight (ELBW) infants. For infants included in the NICHD Neonatal Research Network Generic Database whose mothers were given prenatal MgSO4, data were prospectively collected on maternal/infant conditions and magnesium exposure (including indications, timing and duration of exposure).

DETAILED DESCRIPTION:
Retrospective studies suggested that the risk of cerebral palsy and intraventricular hemorrhage (IVH) in extremely premature infants of mothers given magnesium sulfate (MgSO4) may be reduced. The purpose of this study was to examine the effects of MgSO4 exposure on adverse outcomes in extremely low birth weight (ELBW) infants. For infants included in the NICHD Neonatal Research Network Generic Database, data were prospectively collected on maternal/infant conditions and MgSO4 exposure (including indications, timing and duration of exposure).

ELIGIBILITY:
Inclusion Criteria:

* Infants born in NRN Centers with a birth weight of 401-1,500g

Exclusion Criteria:

* None

Max Age: 14 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: All infants with birth weights 401 through 1500 grams admitted to the NICU within 14 days of age are eligible for the study. In addition, all inborn, liveborn infants in the same weight range (401-1500 gms) who die prior to admission to the NICU are enrolled posthumously.
Sampling Method: Probability Sample
Enrollment: 1339 (Actual)
Dates: Start 1996-07; Primary Completion 1998-06 (Actual); Study Completion 2000-06 (Actual)

PRIMARY OUTCOMES:
Incidence of Intraventricular Hemorrhage | Hospital discharge 120 days of life

SECONDARY OUTCOMES:
Incidence of cerebral palsy | 18-22 months corrected age

CONTACTS AND LOCATIONS:
Overall Officials: James A. Lemons, MD, Study Director — Indiana University; Waldemar A. Carlo, MD, Principal Investigator — University of Alabama at Birmingham; William Oh, MD, Principal Investigator — Brown University, Womens and Infants Hospital; Avroy A. Fanaroff, MD, Principal Investigator — Case Western Reserve University, Rainbow Babies & Children's Hospital; Edward F. Donovan, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati; Barbara J. Stoll, MD, Principal Investigator — Emory University; Ann R. Stark, MD, Principal Investigator — Brigham and Women's Hospital; Charles R. Bauer, MD, Principal Investigator — University of Miami; Lu-Ann Papile, MD, Principal Investigator — University of New Mexico; David K. Stevenson, MD, Principal Investigator — Stanford University; Sheldon B. Korones, MD, Principal Investigator — University of Tennessee; Jon E. Tyson, MD MPH, Principal Investigator — University of Texas Southwestern Medical Center; Seetha Shankaran, MD, Principal Investigator — Wayne State University; Richard A. Ehrenkranz, MD, Principal Investigator — Yale University; Raymond Bain, PhD, Principal Investigator — George Washington University
Locations (15):
- United States (15):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Stanford University, Palo Alto, California
  - Yale University, New Haven, Connecticut
  - George Washington University, Washington D.C., District of Columbia
  - University of Miami, Miami, Florida
  - Emory University, Atlanta, Georgia
  - Indiana University, Indianapolis, Indiana
  - Harvard University, Cambridge, Massachusetts
  - Wayne State University, Detroit, Michigan
  - University of New Mexico, Albuquerque, New Mexico
  - Cincinnati Children's Medical Center, Cincinnati, Ohio
  - Case Western Reserve University, Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - Brown University, Women & Infants Hospital of Rhode Island, Providence, Rhode Island
  - University of Tennessee, Memphis, Tennessee
  - University of Texas Southwestern Medical Center at Dallas, Dallas, Texas

REFERENCES:
- See also: NICHD Neonatal Research Network — http://neonatal.rti.org/